CLINICAL TRIAL: NCT06493045
Title: A Prospective, Single-centre, Randomised, Double-blind, Placebo-controlled, Phase I, First-In-Human (FIH) Trial Evaluating the Safety and Tolerability of Single and Multiple Ascending Oral Doses of IRL757 in Healthy Volunteers
Brief Title: First-In-Human (FIH) Trial Evaluating the Safety and Tolerability of Single and Multiple Ascending Oral Doses of IRL757 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRL757C001
Record Dates: First submitted 2024-05-29; First posted 2024-07-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Not Determined

STUDY DESIGN:
Intervention Model Description: Ascending doses
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IRL757 (Experimental)
  Interventions: Drug: IRL757
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IRL757 — IRL757 capsule
  Arms: IRL757
Drug: Placebo — Placebo capsule
  Arms: Placebo Comparator

SUMMARY:
This is a Phase 1, First-In-Human study evaluating the safety and tolerability of single and multiple ascending oral doses of IRL757 in healthy volunteers.

DETAILED DESCRIPTION:
The trial is composed of two parts: Single Ascending Dose (SAD) part and Multiple Ascending Dose (MAD) part.

The SAD part of the trial will be a parallel group design with one pre-defined starting dose and up to four tentative ascending dose levels of IRL757. Eligible and consenting participants will be included in one of five cohorts, with 8 participants in each cohort (ratio 1:3 placebo/IRL757).

The MAD part of the trial will start after completion of the SAD part of the trial. Depending on the data from the SAD part, two or three dose levels will be evaluated in the MAD part of the trial. There will be 12 participants in each cohort (ratio 1:3 placebo/IRL757).

At the screening visit, consenting subjects will be screened for eligibility according to study specific inclusion/exclusion criteria within 4 weeks before Investigational Medicinal Product (IMP) administration.

If eligible, participants will be admitted to the phase 1 clinic for allocation and administration of the IMP: single dose in the SAD part of the trial or repeated dose (treatment administered repeatedly for 10 days) in the MAD part of the trial. Participants will receive IRL757 or placebo, as randomized.

The treatment allocation will be double-blind, i.e. it will not be disclosed to the patients, the site staff or the Sponsor.

A follow-up visit will be performed for all participants, 5-10 days after IMP administration.

Safety assessments will be performed throughout the study: review and collection of adverse events, physical examination, suicidality ideation, electrocardiogram recording, vital signs, safety laboratory assessments. Blood and urine sampling will also be performed for determination of pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Healthy male or female subject aged 18-55 years inclusive.
* Weight of at least 50 kg and no more than 110 kg at screening.
* Willing to use highly effective methods of contraception

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the trial, or influence the results or the subject's ability to participate in the trial.
* History or present clinically significant psychiatric diagnosis, at discretion of the Investigator.
* Any suicidal ideation of type 4 or 5 in the C-SSRS in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
* History of seizures, including febrile seizure in childhood.
* Any clinically significant illness, medical/surgical procedure or trauma within four (4) weeks of the first administration of IMP.
* Any planned major surgery within the duration of the trial.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
* After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges: Systolic blood pressure > 140 mm Hg, Diastolic blood pressure > 90 mm Hg, Heart rate < 40 or > 85 beats per minute.
* Prolonged QTcF (> 450 ms for male subjects or > 470 ms for female subjects), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
* History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to IRL757.
* Use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two (2) weeks prior to the first administration of IMP, except occasional intake of paracetamol (maximum 2 000 mg/day; and not exceeding 3 000 mg/week), at the discretion of the Investigator.
* Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical trial that included drug treatment within three (3) months of the first administration of IMP in this trial. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
* Current smokers or users of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three (3) times per week is allowed before screening visit.
* History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
* Positive screen for drugs of abuse at screening or on admission to the unit or positive screen for alcohol at screening or on admission to the unit prior to administration of the IMP.
* Use of anabolic steroids.
* Current excessive use of caffeine, as judged by the Investigator.
* Plasma donation within one (1) month of screening or any blood donation/blood loss > 450 mL during the three (3) months prior to screening.
* Investigator considers the subject unlikely to comply with trial procedures, restrictions and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of frequency, seriousness and intensity of adverse events | Until 5-10 days after IMP administration
Description of physical examination findings | Until 5-10 days after IMP administration
Description of electrocardiogram findings | Until 5-10 days after IMP administration
Description of vital signs findings | Until 5-10 days after IMP administration
Description of safety laboratory measurements | Until 5-10 days after IMP administration
Description of C-SSRS (Columbia Suicide Severity Rating Scale) findings | Until 5-10 days after IMP administration

SECONDARY OUTCOMES:
Determination of Maximum Plasma Concentration [Cmax] of IRL757 and its 3 main metabolites | Until 48 hours post-dose
Determination of the AUC of IRL757 and its 3 main metabolites after single and multiple dose | Until 48 hours post-dose
Determination of the time for maximum concentration [Tmax] of IRL757 and its 3 main metabolites | Until 48 hours post-dose
Determination of the half-life [t1/2] of IRL757 and its 3 main metabolites | Until 48 hours post-dose
Determination of the renal clearance (CLr) of IRL757 and its 3 main metabolites | Until 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No